CLINICAL TRIAL: NCT01565564
Title: A Randomized Translational Study to Examine the Effects of Shared Care Versus Usual Care in Management of Gestational Diabetes in a Three-tier Prenatal Care Network in Tianjin, China
Brief Title: Randomized Translational Study to Examine the Effects of Shared Care in Management of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Women and Children's Health Center (Other)
Collaborators: Tianjin Medical University (Other); Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009-02
Record Dates: First submitted 2012-03-21; First posted 2012-03-28 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus; intervention; shared care; pregnancy outcome; macrosomia; pregnancy-induced hypertension
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The usual care arm (Active Comparator)
  Interventions: Behavioral: Shared glycaemic control care within the local three-tier's antenatal care network
- The shared care arm (Active Comparator)
  Interventions: Behavioral: Shared glycaemic control care within the local three-tier's antenatal care network

INTERVENTIONS:
Behavioral: Shared glycaemic control care within the local three-tier's antenatal care network — * Individualized dietary and physical activity consultation plus group diabetes education
  * Self blood glucose monitoring
  * Insulin therapy if indicated
  * Self blood glucose monitoring
  * Insulin therapy institutions if indicated;
  Other Names: The shared lifestyle intervention arm

SUMMARY:
Research question (s)/hypothesis:

1. . The effectiveness of the shared care management of gestational diabetes mellitus;
2. . The cost-effectiveness of the shared care management;
3. . Its sustainability

DETAILED DESCRIPTION:
Method (s) Tianjin three-tier antenatal care network established a universal screening program for gestational diabetes mellitus (GDM) in 1998 and up to 2008, the screening program had screened 115348 pregnant women. GDM will be defined as either fasting plasma glucose (PG) ≥5.1 mmol/L or 1-hour PG≥ 10.0 mmol/L or 2-hour PG≥ 8.5 mmol/L after 75 g glucose tolerance test. A total of 920 pregnant women who have GDM and agree to participate will be randomly assign to have the shared care (diet, physical activity and insulin if indicated) or the local usual antenatal care. The sample size has ≥80% power at a 5% type I error to detect the difference in the primary endpoint, birth weight ≥4000 gram and the secondary endpoint, pregnancy-induced hypertension. Hyperglycemia and other clinical data in the two groups of women will be collected during the shared care or the usual care. Logistic regression and cost-effectiveness analysis will be used in the data analysis.

Public health significance: The introduction of the proven management of GDM in Tianjin antenatal care network will justify the universal screening for GDM and reduce the rate of macrosomic infants and reduce pregnancy-induced hypertension, and thus improve pregnancy outcomes of women with GDM.

Sustainability plan: Just as the universal GDM screening in 1998, the shared care model will be introduced into the Tianjin antenatal care network as part of the usual care routine after the proposed study. The success of the care model will also be publicized and expanded to suburban districts and rural counties of Tianjin, possibly other parts of world where universal screening for GDM is a routine practice.

ACKNOWLEDGEMENT This project is supported by a BRIDGES grant from the International Diabetes Federation. BRIDGES, an International Diabetes Federation project, is supported by an educational grant from Lilly Diabetes."

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who are diagnosed to have GDM.

Exclusion Criteria:

* Diagnosis of overt diabetes during OGTT;
* Younger than 18 years of age;
* Non-singleton pregnancy;
* Maternal-foetal ABO blood type incompatibility;
* Maternal diseases such as chronic hypertension,thyrotoxicosis, prepregnancy diabetes and use of long-term medications that may affect glucose metabolism.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 948 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gongshu Liu, MD, Study Chair — Women and Children's Health Center
Locations (1):
- Tianjin Women and Children's Health Center, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Li J, Liu J, Zhang C, Liu G, Leng J, Wang L, Li W, Yu Z, Hu G, Chan JCN, Yang X. Effects of Lifestyle Intervention of Maternal Gestational Diabetes Mellitus on Offspring Growth Pattern Before Two Years of Age. Diabetes Care. 2021 Mar;44(3):e42-e44. doi: 10.2337/dc20-2750. Epub 2021 Jan 25. No abstract available. PMID 33495293
- [Derived] Yang X, Tian H, Zhang F, Zhang C, Li Y, Leng J, Wang L, Liu G, Dong L, Yu Z, Hu G, Chan JC. A randomised translational trial of lifestyle intervention using a 3-tier shared care approach on pregnancy outcomes in Chinese women with gestational diabetes mellitus but without diabetes. J Transl Med. 2014 Oct 28;12:290. doi: 10.1186/s12967-014-0290-2. PMID 25349017

RESULTS

PARTICIPANT FLOW:
Groups:
- The Shared Care Arm; The Usual Care Arm: Shared glycaemic control care within the local three-tier's antenatal care network: ·Individualized dietary and physical activity consultation plus group diabetes education
  * Self blood glucose monitoring
  * Insulin therapy if indicated
  * Self blood glucose monitoring
  * Insulin therapy institutions if indicated;
Period: Overall Study
Arm/Group | The Shared Care Arm | The Usual Care Arm
Started | 344 | 362
Completed | 339 | 361
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Usual Care Arm | The Shared Care Arm | Total
Number analyzed (Participants) | 361 | 339 | 700
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (3.2) | 29.9 (3.5) | 29.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 339 | 700
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 361 | 339 | 700
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 361 | 339 | 700
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 361 | 339 | 700
Region of Enrollment [Number; unit: participants]
  China | 361 | 339 | 700

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Macrosomia.
Description: Macrosomia is defined as birthweight ≥ 4000 gram.
Time Frame: At the time of birth.
Measure: Number; unit: participants
Arm/Group | The Usual Care Arm | The Shared Care Arm
Number analyzed (Participants) | 361 | 339
participants | 63 | 38

2. Secondary Outcome: The Rate of Pregnancy-induced Hypertension.
Description: Pregnancy-induced hypertension includes gestational hypertension and preeclampsia/eclampsia.
Time Frame: From enrolment at 24-28 gestational weeks till after delivery, an average of 12 weeks.
Measure: Number; unit: participants
Arm/Group | The Usual Care Arm | The Shared Care Arm
Number analyzed (Participants) | 361 | 339
participants | 16 | 27

ADVERSE EVENTS:
Arm/Group | The Shared Care Arm | The Usual Care Arm
Serious Adverse Events (participants affected / at risk) | 0/361 | 0/339
Other Adverse Events (participants affected / at risk) | 0/361 | 0/339

LIMITATIONS AND CAVEATS:
Exclusion of 242 women with GDM diagnosed from 10 Nov 2011 to 31 Jul 2012 due to potential contaminations due to logistic reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No